CLINICAL TRIAL: NCT02938078
Title: Ocular Comfort and Markers of Inflammation in Subjects Undergoing Lid Hygiene Therapy
Brief Title: Ocular Comfort and Inflammation in Lid Hygiene Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota Eye Consultants, P.A. (Industry)
Collaborators: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC-NBY-2016
Record Dates: First submitted 2016-10-14; First posted 2016-10-19 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Eye (Experimental): One eye will be treated with Avenova; the other eye will not be treated. The investigator is masked as to which eye is receiving Avenova product.
  Interventions: Device: Avenova Lid Cleanser
- Non-Treatment Eye (No Intervention): One eye will be treated with Avenova; the other eye will not will be treated. The investigator is masked as to which eye is receiving Avenova product.

INTERVENTIONS:
Device: Avenova Lid Cleanser — Avenova lid cleanser is an FDA-cleared saline solution preserved with 0.01% pure hypochlorous acid.
  Arms: Treatment Eye

SUMMARY:
The primary study objectives are: to evaluate (1) the change in ocular discomfort at 30 days and (2) the change in signs and symptoms of ocular surface disease in demodex-positive subjects beginning the use of Avenova.

DETAILED DESCRIPTION:
This is a prospective study of subjects who have been diagnosed with bilateral demodex blepharitis. Qualified symptomatic eyes will be randomized and monitored for 30 days; one eye will undergo Avenova treatment twice daily and one eye will not undergo any study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed and dated a IRB-approved informed consent document
* Mild or greater Demodex (minimum 15 observable mites in six lashes)
* Score of 20 or more on the OSDI Questionnaire
* Score of 20 or more on the Eyelid Inflammation Questionnaire

Exclusion Criteria:

* Currently enrolled in another prospective research study
* Unable to attend two follow-up visits over 30 days
* Current allergic conjunctivitis of the cornea, conjunctiva, or eyelid in either eye
* Prior ocular trauma where surgery was indicated
* Prior corneal transplant in either eye
* Any ocular surgery within the past six months
* Abnormal corneal scarring, erosions, or Stevens-Johnson syndrome
* Anticipation of ocular surgery within the next 30 days
* Non-English speaking
* Pregnant, nursing, or expect to become pregnant within the next 30 days
* Known sensitivity to chlorine or Avenova
* Moderate, or severe conjunctivochalasis
* Contact lenses within the last 30 days and unwilling to discontinue for 30 days
* Use of topical cyclosporine for less than 6 continuous months prior to baseline
* Procedure such as pulsed light or commercial lid massage in last 30 days
* Known history of autoimmune disease
* Punctal plugs placed within the last 30 days
* Use of Avenova or other lid cleansers within the last 30 days
* Changes in systemic or ocular medications in the last 30 days
* Unwilling to commit to the same ocular and systemic medications for 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Change in Severity of Markers of Inflammation | 30 days
  Clinical parameters include prevalence of demodex mites.
Change in Severity of Markers of Inflammation | 30 days
  Clinical exam parameters include prevalence of tear film break up time.
Change in Severity of Markers of Inflammation | 30 days
  Clinical exam parameters include corneal and conjunctival staining.
Change in Severity of Markers of Inflammation | 30 days
  Clinical parameters include evaluation of meibomian gland including evaluation of lipid layer thickness..
Change in Severity of Markers of Inflammation using tear osmolarity. | 30 days
  Clinical parameters include tear osmolarity.
Change in Severity of Markers of Inflammation | 30 days
  Clinical parameters include tear ferning patterns.
Change in Severity of Markers of Inflammation | 30 days
  Clinical parameters include meibomian gland evaluation
Change in Ocular Discomfort | 30 days
  Change in ocular discomfort based on scores from Eyelid Inflammation questionnaire.
Change in Ocular Discomfort | 30 days
  Change in ocular discomfort based on scores from Ocular Surface Disease Index questionnaire. Scored on a scale of 0-100, with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Fahmy, OD, Principal Investigator — Minnesota Eye Consultants
Locations (1):
- Minnesota eye Consultants, PA, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No